CLINICAL TRIAL: NCT06415058
Title: A Prospective, Nonrandomized Controlled Clinical Investigation of Blood Samples Drawn With the HEMOIV System During Continuous IV Flow
Brief Title: Study to Investigate Blood Samples Drawn With the HemoIV System
Status: Terminated | Type: Observational
Why Stopped: Enrollment limitation
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: MedTG LLC (Unknown)
Responsible Party: Principal Investigator, Brian Bales, Associate Professor, Emergency Medicine, Vanderbilt University Medical Center
Other Study IDs: HemoIV
Record Dates: First submitted 2024-05-01; First posted 2024-05-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Measurement of Blood Parameter Equivalency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- HemoIV Blood Sampling: Measurement of protocol specified blood parameters drawn from the HemoIV system
  Interventions: Device: HemoIV
- Control Blood Sampling: Measurement of protocol specified blood parameters drawn from the contralateral control arm

INTERVENTIONS:
Device: HemoIV — A sterile, single use device. It is a non-patient stick blood collection device that attaches to a peripheral IV catheter (PIV catheter) and allows for blood sample collection to occur during continuous IV infusion therapy. The control blood sampling will occur via standard of care blood draws either through peripheral IV catheter or standard venipuncture.
  Groups: HemoIV Blood Sampling

SUMMARY:
The goal of this study is to compare blood drawn using a device called HemoIV to standard-of-care blood drawn from a vein in the arm or from an IV catheter. The HemoIV is a device that is attached to an IV line. This device allows for blood to be drawn while a patient is receiving IV fluids.

The main questions it aims to answer are:

* Will the HemoIV device allow blood to be drawn without having to stop IV fluids?
* Will the HemoIV device provide the same laboratory results as blood draws done by current standard practice?

Participants will:

* Receive standard medical procedures and/or treatment;
* Have a HemoIV device inserted into their IV line in one arm;
* Have an blood drawn twice from the HemoIV and from an IV line or needle stick from a vein in the other arm. The second blood draw will be done about 8-22 hours after the first blood draw;
* Have the device removed after the second blood draw;
* Receive a phone call about 8 days later to see how you are doing.

DETAILED DESCRIPTION:
The HemoIV investigational device allows for continuous administration of intravenous fluids for blood draw sampling without exposing patients to additional needle sticks, stoppage of intravenous therapy, and potential exposure to bacteria that are inherent risks when performing blood draws using traditional phlebotomy methods. The purpose of this study is to demonstrate the safety and effectiveness of the HemoIV system.

Participants serve as their own control to compare blood measurement parameters. Blood measurements extracted from the participant will be used to compare the control blood sample(s) to the HemoIV blood sample(s). The contralateral arm to the placement of the HemoIV will be the control arm of the study. It is hypothesized that the HemoIV will provide blood samples within the equivalency margin, compared to standard practice (Venipuncture or Peripheral IV Catheter).

The main objectives are:

* To quantitatively measure and compare blood samples drawn with the HemoIV system during continuous intravenous infusion to blood samples from the contralateral arm to demonstrate safety and efficacy of the HemoIV system
* To quantitatively measure and compare the potential advantages of HemoIV to Venipuncture or Peripheral IV Catheter blood draws

Participant population will consist of adult patients admitted to the hospital for a medical condition in the emergency department, inpatient, or observation units and are requiring blood draws as well as intravenous fluids.

Participants will:

* Receive standard of care intravenous therapy via HemoIV inserted through an established peripheral IV catheter
* Have blood samples obtained twice over a 24 hour period from the HemoIV and from an IV line or standard venipuncture from the contralateral arm
* The second blood sampling will occur approximately 8-22 hours after the first blood sampling
* The HemoIV device will be removed one hour after the second blood sampling occurs
* Participants will be called 8 days later to assess for adverse events

Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 and older
* Willing to adhere to the HemoIV intervention regimen
* Patient scheduled for a hospital procedure for medical condition requiring peripheral intravenous catheter placement, intravenous therapy, and blood draw
* Patients to receive intravenous therapy including: Normal Saline, Lactate Ringer, or 5% Dextrose in Water.
* Patient with peripheral intravenous catheter access vein size > 2 mm in diameter or per investigator discretion able to accept an 18G Peripheral Intravenous Catheter.
* Patient must be able to have a peripheral IV catheter in one arm and can have standard venipuncture blood draws from contralateral arm.
* Patient must be able to have an 18G Peripheral Intravenous Catheter inserted for use with the study device up to 1.88" in length.

Exclusion Criteria:

* Do not speak/understand English
* Patients who have a prior history of mastectomy
* Concurrent participation/treatment with another investigational drug or other intervention study.
* Patient with signs and symptoms of thrombophlebitis at the IV site at the time of study enrollment
* Patients receiving chemotherapy, or who have leukemia for example who have fragile formed cellular element
* Patients which are hemodynamically unstable
* Patients requiring blood transfusion via the 18G peripheral IV catheter used with HemoIV
* Patients who are unable to have a peripheral IV catheter on one upper extremity while having the other upper extremity available for blood tests (e.g. subjects must have two arms, not have an AV graft or fistula anticipating dialysis in the near future, etc.)
* Subjects who are not able to have an IV infusion rate adjusted in the HemoIV to between 10-250 mL/hr during blood draws via HemoIV
* Patient with morbid obesity, (BMI > 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient population will be enrolled from those admitted in the hospital (emergency department, inpatient, and observation setting) for a medical condition that require peripheral intravenous catheter fluids and blood draws up to a 24 hour period. Patients receiving Normal Saline, Lactate Ringer, or 5% Dextrose in Water will be enrolled.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Measurement of Whole Blood Count (WBC) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  White Blood Cell Count (WBC) Min: 3.9 to Max:10.7 (10 to the power of 3/uL)
Measurement of Red Blood Count (RBC) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Red Blood Cell Count (RBC) Min: 4.0 to Max: 6.0 (10 to the power of 6/uL)
Measurement of Hemoglobin (HGB) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Hemoglobin (HGB) Min: 11.8 to Max: 18.1 g/dl
Measurement of Hematocrit (HCT) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Hematocrit (HCT) Min: 36% to Max: 49%
Measurement of Platelets (PLT) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Platelets (PLT) Min: 135 to Max: 371 (10 to the power of 3/uL)
Measurement of Albumin (ALB) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Albumin (ALB) Min: 3.2 to Max: 5.2 g/dL
Measurement of Alkaline Phosphatase (AKP) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Alkaline Phosphatase (AKP) Min: 40 to Max: 164 u/L
Measurement of Total Bilirubin (T BILI) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Total Bilirubin (T BILI) Min: 0.1 to Max: 1.2 mg/dL
Measurement of Bicarbonate (CO2) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Bicarbonate (CO2) Min: 17 to Max: 31 mmol/L
Measurement of Blood Urea Nitrogen (BUN) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Blood Urea Nitrogen (BUN) Min: 7 to Max: 26 mg/dL
Measurement of Calcium (CA) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Calcium (CA) Min: 8.4 to Max: 10.5 mg/dL
Measurement of Chloride (CL) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Chloride (CL) Min: 98 to Max: 107 mmol/L
Measurement of Creatinine (Cr) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Creatinine (Cr) Min: 0.57 to Max: 1.25 mg/dL
Measurement of Glucose (Glu) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Glucose (Glu) Min: 70 to Max: 99 mg/dL
Measurement of Potassium (K) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Potassium (K) Min: 3.3 to Max: 4.8 mmol/L
Measurement of Total Protein (TP) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Total Protein (TP) Min: 6.0 to Max: 8.3 g/dL
Measurement of Aspartate Aminotransferase (AST) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Aspartate Aminotransferase (AST) Min: 5 to Max: 35 u/L
Measurement of Alanine Transaminase (ALT) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Alanine Transaminase (ALT) Min: 0 to Max: 55 u/L
Measurement of Sodium (NA) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Sodium (NA) Min: 136 to Max: 145 mmol/L
Measurement of Lactate Dehydrogenase (LDH) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Lactate Dehydrogenase (LDH) Min: 125 to Max: 250 u/L
Measurement of International normalized ratio (INR)/ Prothrombin Time (PT) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  International normalized ratio (INR)/ Prothrombin Time (PT) Min: 11.7 to Max: 14.5 seconds
Measurement of Partial Thromboplastin Time (PTT) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Partial Thromboplastin Time (PTT) Min: 23.5 to Max: 35.5 seconds
Measurement of Fibrinogen parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Fibrinogen Min: 220 to Max: 415 mg/dL
Measurement of Total Cholesterol (CHOL) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Total Cholesterol (CHOL) Min: 0 to Max: 199 mg/dL
Measurement of Triglycerides (TRIG) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Triglycerides (TRIG) Min: 0 to Max: 149 mg/dL
Measurement of High Density Lipoprotein (HDL) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  High Density Lipoprotein (HDL) Min: 0 to Max: 100 mg/dL
Measurement of Low Density Lipoprotein (LDL) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Low Density Lipoprotein (LDL) Min: 0 to Max: 300 mg/dL
Measurement of Troponin I parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Troponin I Min: 0.00 to Max: 0.03 ng/mL
Measurement of Natriuretic Peptides (BNP) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Natriuretic Peptides (BNP) Min: 10 to Max: 100 pg/mL
Measurement of C-Reactive Protein (CRP) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  C-Reactive Protein (CRP) Min: 0 to Max: 5 mg/dL
Measurement of Erythrocyte Sedimentation Rate (ESR) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Erythrocyte Sedimentation Rate (ESR) Min: 1 to Max: 37 mm/hr
Measurement of Human chorionic gonadotropin (HCG) parameter equivalency with HemoIV to the control arm standard of care phlebotomy techniques. | Time point 0 hour (at time of device insertion) and 8-22 hour (post device insertion)
  Human chorionic gonadotropin (HCG) Min: 0 to Max: 5 mIU/mL

SECONDARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale. | Timepoint 0 hour (at time of device insertion) and 8-22 hours (post device insertion)
  Wong-Baker Faces Pain Rating Scale is a method for someone to self-assess and effectively communicate the severity of pain they may be experiencing. The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst."
Study staff usability evaluation of the insertion of HemoIV device. | Timepoint 0 hour (at time of device insertion) and 8-22 hours (post device insertion)
  Study staff will rate the insertion of the device using a difficulty scale from 1-5. 1=Very Difficult, 2= Difficult, 3=Neutral, 4=Easy, 5=Very Easy
Study staff usability evaluation of blood sample collection from the HemoIV device. | Timepoint 0 hour (at time of device insertion) and 8-22 hours (post device insertion)
  Study staff will rate the blood sample collection from the HemoIV device using a difficulty scale from 1-5. 1=Very Difficult, 2= Difficult, 3=Neutral, 4=Easy, 5=Very Easy
Study staff usability evaluation of the ease of the IV solution infusion with the HemoIV device. | Timepoint 0 hour (at time of device insertion) and 8-22 hours (post device insertion)
  Study staff will rate the easy of the IV solution infusion with the HemoIV using a difficulty scale from 1-5. 1=Very Difficult, 2= Difficult, 3=Neutral, 4=Easy, 5=Very Easy
Study staff usability evaluation of the easy of the clearing of the blood channel with the HemoIV device | Timepoint 0 hour (at time of device insertion) and 8-22 hours (post device insertion)
  Study staff will rate the easy of the clearing of the blood channel with the HemoIV using a difficulty scale from 1-5. 1=Very Difficult, 2= Difficult, 3=Neutral, 4=Easy, 5=Very Easy
Study staff usability evaluation of the easy of withdrawal of the HemoIV device | Timepoint 0 hour (at time of device insertion) and 8-22 hours (post device insertion)
  Study staff will rate the easy of withdrawal of the HemoIV using a difficulty scale from 1-5. 1=Very Difficult, 2= Difficult, 3=Neutral, 4=Easy, 5=Very Easy

CONTACTS AND LOCATIONS:
Overall Officials: Sean Collins, MD, MSCi, Study Director — Vanderbilt University Medical Center; Brian Bales, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No